CLINICAL TRIAL: NCT07107308
Title: Efficacy and Safety Evaluation of Microfocused Ultrasound Combined With 1550 nm Non-Ablative Fractional Laser for Facial Rejuvenation: A Randomized, Self-Controlled Clinical Study
Brief Title: Efficacy and Safety Evaluation of Microfocused Ultrasound Combined With 1550 nm Non-Ablative Fractional Laser for Facial Rejuvenation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Weihui Zeng, Professor, Second Affiliated Hospital of Xi'an Jiaotong University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2025008
Record Dates: First submitted 2025-06-03; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Photo-aged Skin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Microfocused Ultrasound Device (MFUpro, Zhengzhou, China) (Experimental)
  Interventions: Device: Microfocused Ultrasound
- Erbium-Doped Fiber Laser Therapeutic Device(FraxStar ShenGuang 1550, Beijing, China) (Experimental)
  Interventions: Device: Erbium-Doped Fiber Laser

INTERVENTIONS:
Device: Microfocused Ultrasound — Before treatment, clean the treatment area, mark the treatment zone, and evenly apply a layer of ultrasound coupling agent about the thickness of a coin on the treatment area. The patient's face was treated with S1.5, S2, N3, N4.5, P1.5, P2.0, P3.0 and P4.5 treatment heads respectively. After the treatment, the face was cleaned and a medical mask was applied for 15 minutes. After the treatment, attention was paid to moisturizing and sun protection.
  Arms: Microfocused Ultrasound Device (MFUpro, Zhengzhou, China)
Device: Erbium-Doped Fiber Laser — Doctors and patients wear corresponding protective glasses. Apply cold gel to the treatment area on the patient's face and select certain treatment parameters based on the patient's skin lesion condition and skin type. After the treatment, clean your face. Decide whether to apply ice based on the severity of the skin lesion reaction. If ice application is necessary, the regular ice application time is 15 to 30 minutes, and apply a medical mask for 15 minutes. After the treatment, pay attention to moisturizing and sun protection.
  Arms: Erbium-Doped Fiber Laser Therapeutic Device(FraxStar ShenGuang 1550, Beijing, China)

SUMMARY:
This study adopted the research method of a single-center case-control study. According to the inclusion and exclusion criteria, 25 patients with facial photoaging were included. After the treatment, various skin indicators of the patients were evaluated and followed up.

Both the researchers and the subjects were in an open state. The researchers measured and evaluated various indicators of the patients' skin. Patients diagnosed with facial photoaging underwent VISIA photography, digital camera photography, non-invasive skin testing, dermoscopy testing and high-frequency skin ultrasound testing after enrollment. On the day of enrollment, micro-focused ultrasound (using treatment heads S1.5, S2, N3, N4.5, P1.5, P2.0, P3.0, and P4.5) was performed on both sides of the face once. One side of the face was randomly selected as the experimental side, and a 1550 nm non-ablative fractional laser treatment was performed immediately after the micro-focused ultrasound treatment once. For the second treatment, micro-focused ultrasound (using S1.5, S2, P1.5, and P2.0 treatment heads) was performed on both sides once. The experimental side was treated with 1550 nm non-ablative fractional laser once immediately after the micro-focused ultrasound treatment.

The research period was May, including a treatment period of 2 months. Follow-up was conducted every two weeks for a total of 10 times, all of which were on-site visits. The grace period during the visit is ±3 days.

DETAILED DESCRIPTION:
This study intends to perform micro-focused ultrasound combined with 1550nm non-ablative fractional laser treatment on patients with facial photoaging, and evaluate its efficacy and safety for facial photoaging. It aims to observe whether the efficacy of micro-focused ultrasound combined with 1550nm non-ablative fractional laser for facial photoaging is superior to that of micro-focused ultrasound treatment alone.

This study adopted the research method of a single-center case-control study. According to the inclusion and exclusion criteria, 25 patients with facial photoaging were included. The assessment and follow-up of various skin indicators of the patients were conducted before and after the treatment. Both the researchers and the subjects were in an open state. The researchers measured and evaluated various indicators of the patients' skin.

1. Preparatory work: Twenty-five volunteers with photoaging of the skin who met the inclusion criteria were recruited. After the first diagnosis, the informed consent form was signed. The basic information of the patients (age, gender, skin type, nature of work, sun exposure time, expression habits, etc.) was recorded. Digital photos of the front, 45-degree left and right sides, and 90-degree left and right sides were taken manually. The pictures were collected using the VISIA skin detector. The thickness of the dermis at the nasolabial sulcus was measured by skin ultrasound, and dermoscopy was performed. Non-invasive skin physiological indices were measured: skin elasticity, TEWL, EI, MI, and L*a*b* values (the average value was calculated by taking three points from different parts). Meanwhile, the patients underwent self-Rating Anxiety Scale (SAS) and Self-Rating Depression Scale (SDS) scores.
2. Treatment process: Micro-focused ultrasound (using treatment heads S1.5, S2, N3, N4.5, P1.5, P2.0, P3.0, and P4.5) was performed once on both sides of the face. One side of the face was randomly selected as the experimental side. Immediately after the micro-focused ultrasound treatment, a 1550 nm non-ablative fractional laser (with a dot spacing of 0.75-1.25mm) was performed. Energy: 10-20 MJ. Repeat the treatment twice. The endpoint reaction is mild erythema and edema at the treatment site. Treat once. The second treatment was conducted 6 weeks after the first treatment. Micro-focused ultrasound treatment (using S1.5, S2, P1.5, and P2 treatment heads) was performed on both sides once. On the experimental side, 1550 nm non-ablative fractional laser (with a dot spacing of 0.75-1.25mm and an energy of 10-20mj) was performed immediately after micro-focused ultrasound treatment. The treatment was repeated twice. The endpoint response was mild erythema and edema at the treatment site (treated once). A total of 2 treatments were conducted. Use the moisturizing mask continuously for three days after each treatment. After the first diagnosis and the end of follow-up, the patients underwent Self-Rating Anxiety Scale (SAS) and Zong's Self-Rating Depression Scale (SDS) scores. The daily basic care products used by all patients were facial cleanser + simple moisturizer + sunscreen.
3. Follow-up: Follow-up was conducted before each treatment, 2 weeks after the end of the first treatment, 4 weeks after the end of the first treatment, and 2 weeks, 4 weeks, 6 weeks, and 12 weeks after the end of all treatments. During the follow-up, VISIA photography, digital camera photography, dermoscopy detection, high-frequency ultrasound detection of the skin and non-invasive skin detection were performed: skin elasticity, EI, MI, L*a*b* value, TEWL value. Self-rating Anxiety Scale (SAS) and Zong's Self-Rating Depression Scale (SDS) scores were conducted at the end of the first diagnosis and all follow-ups.

Record any adverse events during the trial, any laser and drug adverse reactions, the reasons for withdrawal from the trial, and any clinically significant abnormalities from baseline to the end of follow-up for safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with facial skin photoaging diagnosed by clinicians [Photoaging Score (GPS)1-4 points];
2. Male or female patients aged 30 to 60 years old;
3. Patients with Fitzpatrick9 skin wrinkle grades I to III;
4. Patients who voluntarily participate and sign the informed consent form.

Exclusion Criteria:

1. The degree of photoaging on both sides of the face varies relatively significantly;
2. There are mobile or metal implants on the face;
3. Severe or cystic acne on the face;
4. There was a history of facial injection or surgery within 6 months before the trial;
5. Severe keloid constitution;
6. There is a history of allergy to local anesthetics, iodophor or photosensitivity.
7. Have a history of bleeding tendency;
8. Suffering from serious skin diseases such as skin tumors;
9. Suffering from autoimmune diseases, systemic diseases or mental disorders;
10. Women who are planning to become pregnant, are pregnant or breastfeeding;
11. There is a frequent need for makeup;
12. There is a long-term need for outdoor work and sun protection is not possible.
13. Patients with poor compliance, which affects clinical efficacy and the judgment of adverse reactions.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
GAIS(Global Aesthetic Improvement Scale) Score | week 0、4、8、12、16
  Minimum 0 points, maximum 4 points. The higher the score, the better the therapeutic effect.

SECONDARY OUTCOMES:
Dermal Thickness | week 0、4、8、12、16
  Utilizing the High-frequency Ultrasound Detector

OTHER OUTCOMES:
Melanin Index | week 0、4、8、12、16
  Utilizing the DermaLab® Combo (Cortex Technology)
Erythema Index(EI) | week 0、4、8、12、16
  Utilizing the DermaLab® Combo (Cortex Technology)
Skin Hydration | week 0、4、8、12、16
  Utilizing the DermaLab® Combo (Cortex Technology)
Elasticity Index | week 0、4、8、12、16
  Utilizing the DermaLab® Combo (Cortex Technology)

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hospital of Xi'an Jiaotong University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: No